CLINICAL TRIAL: NCT02869607
Title: Institut Paoli Calmettes Breast Cancer Database
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BDD-SEIN-IPC
Record Dates: First submitted 2016-08-03; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer Diagnosis
MeSH Terms: conditions — Breast Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with breast cancer diagnosis
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
Database of Institut Paoli-Calmettes patients diagnosed with breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of breast cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Breat Cancer
Sampling Method: Non-Probability Sample
Enrollment: 45000 (Estimated)
Dates: Start 1995-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival of patients with breast cancer | 10 years
  Overall survival of all patients who come in the center

SECONDARY OUTCOMES:
Collection of patients characteristics | 10 years
  Collection of characteristics of patients treated at Institut Paoli Calmettes in order to set up prospective and retrospective studies

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houvenaeghel G, de Nonneville A, Cohen M, Sabiani L, Buttarelli M, Charaffe E, Jalaguier A, Bannier M, Tallet A, Viret F, Goncalves A. Neoadjuvant chemotherapy for breast cancer: Pathologic response rates but not tumor size, has an independent prognostic impact on survival. Cancer Med. 2024 Feb;13(3):e6930. doi: 10.1002/cam4.6930. Epub 2024 Feb 7. PMID 38327130
- [Derived] Houvenaeghel G, de Nonneville A, Cohen M, Chopin N, Coutant C, Reyal F, Mazouni C, Gimbergues P, Azuar AS, Chauvet MP, Classe JM, Darai E, Martinez A, Rouzier R, de Lara CT, Lambaudie E, Barrou J, Goncalves A. Lack of prognostic impact of sentinel node micro-metastases in endocrine receptor-positive early breast cancer: results from a large multicenter cohort☆. ESMO Open. 2021 Jun;6(3):100151. doi: 10.1016/j.esmoop.2021.100151. Epub 2021 May 10. PMID 33984674